CLINICAL TRIAL: NCT06788535
Title: A Phase 3, Open-Label, Multicenter Study of I-124 Evuzamitide as an Imaging Agent for the Diagnosis of Cardiac Amyloidosis Using Positron Emission Tomography Computed Tomography (PET/CT)
Brief Title: Research With I-124 EVuzamitide to Elucidate Cardiac AmyLoidosis
Acronym: REVEAL
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sharmila Dorbala (Other)
Collaborators: Attralus, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Sharmila Dorbala, Director Nuclear Cardiology, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024P002136
Record Dates: First submitted 2024-12-23; First posted 2025-01-23 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Cardiac Amyloidosis
Keywords: Amyloid Light Chain (AL); Cardiac Amyloidosis; Amyloidosis; Amyloid Transthyretin (ATTR); Transthyretin (TTR); REVEAL; PET Imaging
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Amyloidosis

STUDY DESIGN:
Masking Description: I-124 evuzamitide PET/CT imaging will be evaluated by three (3) independent readers who are blinded to all clinical data.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single dose, Open label (Experimental): Open label use of I124-evuzamitide to diagnose cardiac amyloidosis.
  Interventions: Drug: I-124 evuzamitide

INTERVENTIONS:
Drug: I-124 evuzamitide — I-124 evuzamitide, single dose imaging agent, administered intravenously.
  Other Names: AT-01

SUMMARY:
The purpose of this Phase 3, open label, single dose imaging study is to evaluate the efficacy and safety of I-124 evuzamitide (radioactive dye) for diagnosing Cardiac Amyloidosis in participants with suspected Cardiac Amyloidosis. The imaging test that will be used in this study is a Positron Emission Tomography Computed Tomography (PET/CT) scan.

DETAILED DESCRIPTION:
This Phase 3, open label, single dose study will evaluate the efficacy and safety of I-124 evuzamitide when administered as a single dose prior to a PET/CT scan. Participants will be in the study for up to 60 days and approximately 200 participants with suspected Cardiac Amyloidosis will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Understands the study procedures and can give signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Male or female ≥18 years of age.
* Is suspected of having cardiac amyloidosis and is undergoing or will undergo a diagnostic evaluation for cardiac amyloidosis (e.g., echocardiography, CMR, bone avid tracer cardiac SPECT, extracardiac or endomyocardial biopsy, etc.). Participants can be enrolled before or during their diagnostic evaluation for cardiac amyloidosis.
* Able to undergo PET/CT imaging as part of the study, including ability to lie supine for approximately 1 hour.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of <1% per year during the treatment period and for at least 30 days after administration of I-124 evuzamitide.
* For men: agreement to remain abstinent or use contraceptive measures and agreement to refrain from donating sperm

Exclusion Criteria:

* Established diagnosis of cardiac amyloidosis.
* Established diagnosis of systemic amyloidosis (e.g., renal AL or ATTR peripheral neuropathy) without known cardiac involvement. Participants who are amyloid positive only with carpal tunnel tissue or laminectomy are allowed as long as they do not have other known organ involvement.
* Receiving therapy with an approved treatment (e.g., tafamadis) or in a clinical trial for treatment for ATTR cardiac amyloidosis at time of enrollment. For AL and ATTR: Patients may enter the screening period of a clinical trial for treatment after the ICF is signed and participant is enrolled in this trial but may not receive an experimental therapy until after the Day 30 safety follow-up visit in this trial.
* Is pregnant or breast-feeding.
* Is mentally or legally incapacitated, has significant emotional problems at the time of the study, or has a history of psychosis.
* Has a known allergy to potassium iodide.
* Receiving hemodialysis or peritoneal dialysis.
* eGFR less than 15mL/min/1.73m2.
* Myocardial infarction within three (3) months of screening.
* Has severe claustrophobia or any condition, medial or otherwise, that would prevent completion of the study assessments.
* Has any illness that, in the opinion of the investigator, might confound the results of the study or pose additional risk to the participant.
* Has received heparin or heparin analogs (e.g., enoxaparin, dalteparin, fondaparinux) within seven (7) days prior to I-124 evuzamitide administration.
* Known uncorrected thyroid disorders (other than mild elevation of thyroid stimulating hormone with normal T4).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2026-02-13 (Estimated); Study Completion 2026-02-13 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of I-124 evuzamitide for diagnosing cardiac amyloidosis-Sensitivity | Up to 60 days after scanning
  Assessment of the sensitivity of PET/CT imaging with I-124 evuzamitide for the diagnosis of cardiac amyloidosis based on visual scan interpretation.
To evaluate the efficacy of I-124 evuzamitide for diagnosing cardiac amyloidosis-Specificity | Up to 60 days after scanning
  Assessment of specificity of PET/CT imaging with I-124 evuzamitide for the diagnosis of cardiac amyloidosis based on visual scan interpretation.

SECONDARY OUTCOMES:
To evaluate the safety of a single intravenous administration of I-124 evuzamitide-Treatment Emergent Adverse Events | 30 days after administration of I-124 evuzamitide
  Incidence of treatment-emergent Adverse Events (AEs) from Day 1 to Day 30.
To evaluate the safety of a single intravenous administration of I-124 evuzamitide-Creatinine | 30 days after administration of I-124 evuzamitide
  Change in kidney function from baseline: Creatinine mg/dl
To evaluate the safety of a single intravenous administration of I-124 evuzamitide-eGFR | 30 days after administration of I-124 evuzamitide
  Change in kidney function from baseline: eGFR ml/min/1.73 m2
To evaluate the safety of a single intravenous administration of I-124 evuzamitide-Liver function. | 30 days after administration of I-124 evuzamitide
  Change in liver function from baseline LDH units per liter; Alkaline phosphatase units per liter; SGOT units per liter; SGPT units per liter
To evaluate the safety of a single intravenous administration of I-124 evuzamitide. | 30 days after administration of I-124 evuzamitide
  Change in pregnancy test from baseline Pregnancy testing beta HCG serum testing negative or positive

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Mayo Clinic, Scottsdale, Arizona
  - City of Hope - Duarte, Duarte, California
  - University of California, San Francisco, California
  - Yale Cardiovascular Medicine, New Haven, Connecticut
  - Cleveland Clinic, Weston, Florida
  - Northwestern University, Chicago, Illinois
  - Cook County Health, Chicago, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - St. Lukes (CVIT) Saint Luke's Health System, Kansas City, Missouri
  - Washington University of St. Louis, St Louis, Missouri
  - Rutgers, New Brunswick, New Jersey
  - Columbia University, New York, New York
  - Duke University, Durham, North Carolina
  - Cone Health, Greensboro, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Houston Methodist, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wall JS, Martin EB, Lands R, Ramchandren R, Stuckey A, Heidel RE, Whittle B, Powell D, Richey T, Williams AD, Foster JS, Guthrie S, Kennel SJ. Cardiac Amyloid Detection by PET/CT Imaging of Iodine (124I) Evuzamitide (124I-p5+14): A Phase 1/2 Study. JACC Cardiovasc Imaging. 2023 Nov;16(11):1433-1448. doi: 10.1016/j.jcmg.2023.08.009. PMID 37940323
- [Result] Clerc OF, Cuddy SAM, Robertson M, Vijayakumar S, Neri JC, Chemburkar V, Kijewski MF, Di Carli MF, Bianchi G, Falk RH, Dorbala S. Cardiac Amyloid Quantification Using 124I-Evuzamitide (124I-P5+14) Versus 18F-Florbetapir: A Pilot PET/CT Study. JACC Cardiovasc Imaging. 2023 Nov;16(11):1419-1432. doi: 10.1016/j.jcmg.2023.07.007. Epub 2023 Sep 6. PMID 37676210